CLINICAL TRIAL: NCT05736367
Title: Pilot Study to Investigate the Metabolic Pathways in Hormone Receptor Positive/HER2 Negative Breast Cancer
Brief Title: Investigating the Metabolic Pathways in Hormone Receptor Positive/HER2 Negative Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Ludwig Institute for Cancer Research (Other)
Responsible Party: Principal Investigator, Coral Omene, Assistant Professor, Medical Oncology, Rutgers Cancer Institute of New Jersey, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 042210; Pro2022002366 (Other: Rutgers, The State University of New Jersey)
Record Dates: First submitted 2023-02-06; First posted 2023-02-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: Hormone Receptor Positive; Metabolic activity; Breast Cancer Surgery; 13C isotope glucose; Metabolomics
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metabolic activity of Hormone Receptor Positive (HR+)/Her 2 Negative (Her2-) Breast cancer (Experimental): Administration of U-13C-glucose to participants with early-stage HR+/Her2- breast cancer fitting criteria, will be done intraoperatively at the time of resection, as well as blood sample collection.
  This will allow for in depth evaluation of glycolysis as well as TCA cycle, lipid and amino acid metabolism and comprehensive genomic analyses to complement the metabolic assays that will be done by the Ludwig Institute of Cancer Research. HR+/Her2- breast cancer subtype is chosen for this feasibility pilot study given that metabolic studies have not been done in this subtype of breast cancer and it makes up the majority of breast cancer cases.
  Interventions: Drug: U-13C-glucose

INTERVENTIONS:
Drug: U-13C-glucose — Discover new insights into the glucose, TCA cycle, amino acid, and lipid metabolic dependencies of HR+/Her2- breast cancer, via liquid chromatography-mass spectrometry (LC-MS) and nuclear magnetic resonance (NMR) spectroscopy analysis of in vivo U-13C-glucose-labeled biopsy of tumor and benign adjacent tissue

SUMMARY:
To analyze the metabolic activity of Hormone Receptor Positive (HR+)/Her 2 Negative (Her2-) Breast cancer.

DETAILED DESCRIPTION:
Participants will be asked to receive a glucose infusion (U-13C- glucose intravenous) during routine breast cancer surgery at which time, tumor biopsy samples and blood samples will be collected to be used in research experiments to help provide insight into the metabolic activity of the tumor. The length of time on study for each patient will be three - four weeks including two to three hours for glucose infusion and breast cancer biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Have hormone receptor (HR) positive [estrogen receptor( ER)+/progesterone receptor (PR)+, ER+/PR- or ER-/PR+)/Her2 negative breast cancer previously diagnosed by biopsy.
* Have early stage, clinical or anatomic stage I, II or III breast cancer (cT1cN0, cT1cN1, cT2N0, cT2N1, cT3N0)
* Candidates for intended curative primary resection who have not had neoadjuvant therapy (endocrine/hormonal therapy, chemotherapy with or without immunotherapy).
* Willing to undergo mandatory intraoperative small excisional and core biopsies (4-6 passes) of tumor and normal tissue for research purposes at the time of proposed surgical resection.

Exclusion Criteria:

* Is currently enrolled, or will enroll in, a different clinical study in which investigational therapeutic procedures are performed or investigational therapies are administered while participating in this study.
* Has triple negative (ER-/PR-/Her2-) or HER2+ breast cancer.
* Concomitant active malignancy
* Is of child-bearing potential who has not had a recent negative pregnancy test done outside of this clinical trial (i.e., as part of standard preparation for diagnosis and treatment for her cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Measure glycolysis metabolism dependencies of hormone receptor positive/HER2 negative breast cancer using Liquid chromatography-mass spectrometry (LC-MS) | Baseline to four weeks
  To analyze and describe the metabolism of these tumors in vivo uniformly-labeled (U-13C)-glucose-labeled biopsy of tumor and benign adjacent tissue. The participants will receive glucose infusion and their tumor specimens analyzed. Blood collection will allow for in depth evaluation of glycolysis metabolism.
  Compounds can range from low molecular mass analytes with m/z values < 1000 Da, to very high molecular mass proteins with m/z values > 100,000 Da
  U-13C-Glucose (study drug)
Measure glycolysis metabolism dependencies of hormone receptor positive/HER2 negative breast cancer using Nuclear Magnetic Resonance (NMR) spectroscopy in parts per million (ppm). | Baseline to four weeks
  To analyze and describe the metabolism of these tumors in vivo uniformly-labeled (U-13C)-glucose-labeled biopsy of tumor and benign adjacent tissue. The participants will receive glucose infusion and their tumor specimens analyzed. Blood collection will allow for in depth evaluation of glycolysis metabolism.
  U-13C-Glucose (study drug)

SECONDARY OUTCOMES:
Measure lipid metabolic dependencies of hormone receptor positive/HER2 negative breast cancer using Liquid chromatography-mass spectrometry (LC-MS) | Baseline to four weeks
  To analyze and describe the metabolism of these tumors in vivo uniformly-labeled (U-13C)-glucose-labeled biopsy of tumor and benign adjacent tissue. The participants will receive glucose infusion and their tumor specimens analyzed. Blood collection will allow for in depth evaluation of lipid metabolism.
Measure lipid metabolic dependencies of hormone receptor positive/HER2 negative breast cancer using Nuclear Magnetic Resonance (NMR) spectroscopy in parts per million (ppm) | Baseline to four weeks
  To analyze and describe the metabolism of these tumors in vivo uniformly-labeled (U-13C)-glucose-labeled biopsy of tumor and benign adjacent tissue. The participants will receive glucose infusion and their tumor specimens analyzed. Blood collection will allow for in depth evaluation of lipid metabolism.
Measure amino acid metabolic dependencies of hormone receptor positive/HER2 negative breast cancer using Liquid chromatography-mass spectrometry (LC-MS). | Baseline to four weeks
  To analyze and describe the metabolism of these tumors in vivo uniformly-labeled (U-13C)-glucose-labeled biopsy of tumor and benign adjacent tissue. The participants will receive glucose infusion and their tumor specimens analyzed. Blood collection will allow for in depth evaluation of amino acid metabolism.
  Compounds can range from low molecular mass analytes with m/z values < 1000 Da, to very high molecular mass proteins with m/z values > 100,000 Da
Measure amino acid metabolic dependencies of hormone receptor positive/HER2 negative breast cancer using Nuclear Magnetic Resonance (NMR) spectroscopy in parts per million (ppm) | Baseline to four weeks
  To analyze and describe the metabolism of these tumors in vivo uniformly-labeled (U-13C)-glucose-labeled biopsy of tumor and benign adjacent tissue. The participants will receive glucose infusion and their tumor specimens analyzed. Blood collection will allow for in depth evaluation of amino acid metabolism.

CONTACTS AND LOCATIONS:
Overall Officials: Coral Omene, MD, PhD, Principal Investigator — Cancer Institute of New Jersey Rutgers
Locations (2):
- United States (2):
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - RWJBarnabas Health, New Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: No